CLINICAL TRIAL: NCT06636903
Title: The Effect of Acupressure Applied Before Suturing Procedure in the Emergency Department on Anxiety and Vital Signs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ezgi BOLAT (Other)
Responsible Party: Sponsor-Investigator, Ezgi BOLAT, graduate student, Mersin University
Organization: Mersin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MU-EBOLAT-804
Record Dates: First submitted 2024-10-01; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Anxiety; Vital Signs
Keywords: Acupressure, Suturing, Anxiety, Vital Signs, Emergency Department
MeSH Terms: conditions — Anxiety Disorders; Emergencies | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Randomized parallel controlled experimental study design
Who Masked: Participant
Masking Description: A biostatistician who is not involved in the study will be randomly assigned to groups A and B created by a biostatistician in a computer environment. As a result of the drawing of lots, whether groups A and B will be the study or control group will be determined by tossing a coin at the beginning of the study. Information indicating that the patients included in the study sample were assigned to groups A and B according to the randomization table will be placed in an opaque envelope. This envelope will be kept by the coordinator researcher (GAU) and when the researcher (EB) goes to the patient for the application, he will open the envelope after filling out the "Informed Consent Form" and learn which group the patient is in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupressure group (Experimental): Acupressure will be applied to the experimental group before suturing.
  Interventions: Other: Acupressure
- control group (No Intervention): No intervention will be made to the control group. Routine emergency room practice will be carried out.

INTERVENTIONS:
Other: Acupressure — Before pressing directly on the point for acupressure, a gentle warming, relaxing and preparatory process of approximately 15 seconds should be performed on the point area. In this case, manual pressure with the thumb, index finger and/or middle finger will be applied sequentially (in the rhythm of breathing) without lifting the finger for an average of 1.5 minutes on each point, at a frequency that does not disturb the person, does not cause pain and has a calming effect. Before the suturing procedure, acupressure will be applied to the HT7 and Li4 points by a researcher (EB) who has an acupressure certificate.
  Arms: Acupressure group
Other: Acupressure — Before and after acupressure, vital signs and before acupressure, anxiety scores will be checked using the Spielger State Anxiety Scale. In addition, vital signs and anxiety scores will be checked again immediately after the stitching procedure.
  Other Names: Acupressure Group
  Arms: Acupressure group

SUMMARY:
This study suggests that the anxiety experienced by patients during suturing in the emergency department can be reduced with acupressure and offers a research proposal on vital signs.

Problem: During suturing in the emergency department, patients experience high levels of anxiety due to the pain they experience and fear of the procedure. This situation complicates the treatment process, negatively affects the health of patients and creates a difficult situation for healthcare professionals.

Solution Suggestion: Acupressure can be used as a non-invasive, safe and effective method to reduce patients' anxiety. Acupressure reduces pain, provides relaxation and reduces anxiety by increasing the secretion of endorphins in the body.

Purpose of the Study: The purpose of this study is to evaluate the effects of applying acupressure to patients before suturing in the emergency department on their anxiety levels and vital signs (such as blood pressure, heart rate).

In summary, this research has a significant potential that emergency room nurses can improve patients' quality of life and make treatment processes more effective by using acupressure in patient care.

Key Words: Acupressure, Suturing, Anxiety, Vital Signs, Emergency Department

ELIGIBILITY:
Inclusion Criteria:

* Suturing is done with local anesthesia,
* Those who are 18 years or older,
* Conscious, oriented and cooperative,
* Able to read and understand Turkish,
* Agreeing to participate in the study,
* Anxiety not diagnosed,
* Not using medication for anxiety,
* No acupressure experience,
* No physical problems that would prevent acupressure application to Ht7 and Li4 points,
* Not pregnant,
* Patients who sign the "Voluntary Informed Consent Form" will be included.

Exclusion Criteria:

* Those who are under 18 years of age,
* Unconscious, unoriented and uncooperative,
* Cannot read and understand Turkish,
* Those who do not agree to participate in the study,
* -Diagnosed with anxiety,
* -Using medication for anxiety (anxiolytic, antidepressant, antipsychotic, etc.),
* Having previous acupressure experience,
* Having a physical problem that prevents the application of acupressure to Ht7 and Li4 points,
* Pregnant,
* Patients who do not sign the "Voluntary Informed Consent Form" will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of anxiety before acupressure | before suturing
  Before the suturing procedure, acupressure will be applied to the Ht7 and Li4 points.The state anxiety scale consists of 20 questions. The statements in the SAS are evaluated as none 1 point, a little 2 points, a lot 3 points and completely 4 points. In this section, the statements are divided into direct and reversed. Reversed statements are: items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20. The SAS score is calculated by adding the constant value of 50 to the value obtained by subtracting the total score of the reversed statements from the total score of the direct statements. The scale score varies between 20-80 and an increase in the score obtained from the scale indicates an increase in the anxiety level. A total score of 0-19 from the SAS indicates no anxiety, a score of 20-39 indicates mild anxiety, a score of 40-59 indicates moderate anxiety and a score of 60-79 indicates a severe anxiety level. It is stated that individuals who score above 60 on the SAS need professional help.
Evaluation of anxiety after suturing | immediately after suturing
  Immediately after the stitching, the anxiety scale will be filled out again. The statements in the SAS are evaluated as none 1 point, a little 2 points, a lot 3 points and completely 4 points. In this section, the statements are divided into direct and reversed. Reversed statements are: items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20. The SAS score is calculated by adding the constant value of 50 to the value obtained by subtracting the total score of the reversed statements from the total score of the direct statements. The scale score varies between 20-80 and an increase in the score obtained from the scale indicates an increase in the anxiety level. A total score of 0-19 from the SAS indicates no anxiety, a score of 20-39 indicates mild anxiety, a score of 40-59 indicates moderate anxiety and a score of 60-79 indicates a severe anxiety level. It is stated that individuals who score above 60 on the DAS need professional help.

SECONDARY OUTCOMES:
Assessment of blood pressure before acupressure | Just before acupressure
  Vital signs will be monitored immediately before acupressure. The patient's blood pressure will be monitored before acupressure. The patients' blood pressure will be monitored on a portable monitor (iMEC 10, Mindray, Chinese). Systolic blood pressure of 100-130 mmHg, diastolic blood pressure of 60-80 mmHg. Normal blood pressure is usually considered to be between 90/60 mmHg and 120/80 mmHg.
Assessment of Blood Pressure After Acupressure | After acupressure
  Vital signs will be monitored immediately after acupressure. The patient's blood pressure will be monitored after acupressure. The patients' blood pressure will be monitored on a portable monitor (iMEC 10, Mindray, Chinese). Systolic blood pressure of 100-130 mmHg, diastolic blood pressure of 60-80 mmHg. Normal blood pressure is usually considered to be between 90/60 mmHg and 120/80 mmHg.
Assesment of blood pressure after suturing | after suturing
  Vital signs will be monitored immediately after suturing. The patient's blood pressure will be monitored after suturing. The patients' blood pressure will be monitored on a portable monitor (iMEC 10, Mindray, Chinese). Systolic blood pressure of 100-130 mmHg, diastolic blood pressure of 60-80 mmHg. Normal blood pressure is usually considered to be between 90/60 mmHg and 120/80 mmHg.
Assesment of heart rate before acupressure | before acupressure
  Vital signs will be monitored immediately before acupressure. The patient's heart rate will be monitored before acupressure. The patient's heart rate will be monitored on a portable monitor (iMEC 10, Mindray, Chinese). A normal heart rate for adults ranges from 60 to 100 beats per minute.
Assesment of heart rate after acupressure | after acupressure
  Vital signs will be monitored immediately after acupressure. The patient's heart rate will be monitored after acupressure. The patient's heart rate will be monitored on a portable monitor (iMEC 10, Mindray, Chinese). A normal heart rate for adults ranges from 60 to 100 beats per minute.
Assesment of heart rate after suturing | after suturing
  Vital signs will be monitored immediately after suturing. The patient's heart rate will be monitored after suturing. The patient's heart rate will be monitored on a portable monitor (iMEC 10, Mindray, Chinese). A normal heart rate for adults ranges from 60 to 100 beats per minute.
Assesment of oxygen saturation before acupressure | before acupressure
  Vital signs will be monitored immediately before acupressure. The patient's heart rate will be monitored before acupressure. The patient's heart rate will be monitored on a portable monitor (iMEC 10, Mindray, Chinese). For most people, a normal pulse oximeter reading for your oxygen saturation level is between 95% and 100%.
Assesment of oxygen saturation after acupressure | after acupressure
  Vital signs will be monitored immediately after acupressure. The patient's heart rate will be monitored after acupressure. The patient's heart rate will be monitored on a portable monitor (iMEC 10, Mindray, Chinese). For most people, a normal pulse oximeter reading for your oxygen saturation level is between 95% and 100%.
Assesment of oxygen saturation after suturing | after suturing
  vVital signs will be monitored immediately after suturing. The patient's heart rate will be monitored after suturing. The patient's heart rate will be monitored on a portable monitor (iMEC 10, Mindray, Chinese). For most people, a normal pulse oximeter reading for your oxygen saturation level is between 95% and 100%.
Assesment of respiratory rate before acupressure | before acupressure
  Immediately before acupressure, the respiratory rate will be assessed. The respiratory rate will be counted by observing the chest cage movements for one minute by the researcher (EB). Vital signs are expected to remain within normal values. Normal respiration rates for an adult person range from 16 to 20 breaths per minute.
Assesment of respiratory rate after acupressure | after acupressure
  Immediately after acupressure, After suturing, the respiratory rate will be assessed. The respiratory rate will be counted by observing the chest cage movements for one minute by the researcher (EB). Vital signs are expected to remain within normal values. Normal respiration rates for an adult person range from 16 to 20 breaths per minute.
Assesment of respiratory rate after suturing | after suturing
  After suturing, the respiratory rate will be assessed. The respiratory rate will be counted by observing the chest cage movements for one minute by the researcher (EB). Vital signs are expected to remain within normal values. Normal respiration rates for an adult person range from 16 to 20 breaths per minute.

IPD SHARING:
Plan to Share IPD: Undecided